CLINICAL TRIAL: NCT06885450
Title: Perforator Pedicled V-Y Advanced Flaps for Coverage of Soft Tissue Defects in the Lower Limbs
Brief Title: Perforator Pedicled V-Y Advanced Flaps for Coverage in the Lower Limbs
Status: Completed | Type: Observational
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: XYFY-SSZX
Record Dates: First submitted 2025-03-11; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Soft Tissue Defects; Perforator Flap
Keywords: the lower leg; soft tissue defects; perforator flaps; dopper ultrasound; advanced flaps

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Perforator Pedicled Flaps — Perforator Pedicled V-Y Advanced Flaps

SUMMARY:
Repair of soft tissue defects with hardware exposing in the lower limbs was considered as a severe challenge for plastic surgeons in reconstructive surgery. The purpose of the paper was to investigate the clinical effect of perforator pedicled V-Y advanced flap for repairing soft tissue defects with hardware exposing in the lower leg .

DETAILED DESCRIPTION:
The various causes of the lower leg defects always consist of trauma, infection, tumors etc. Flaps are often used to cover the wounds when the bones and tendons are exposed to the body surface. However, flap coverage at the lower leg was considered a severe challenge due to the difficult anatomy and paucity of soft tissue1. Reconstruction and esthetic aspects of defect should be systemically considered .Common skin flaps include the peroneal perforator flap, the medial sural artery perforator flap2-8and muscle flaps. However, common skin flaps have a disadvantage of reversing of the pedicle which may be a reason of necrosis. A split thickness skin graft was usually applied to cover close secondary wound at the donor site. The aim of this paper was to investigate the clinical effect of V-Y advanced flaps based on septocutaneous and musculocutaneous perforator in the repair of soft-tissue wounds in the lower limbs.

ELIGIBILITY:
Inclusion Criteria:

1. people age: among 5-80years,
2. tolerate general anesthesia.
3. The perforating vessel is fine.

Exclusion Criteria:

1. patients age :<5years,>80years
2. can not tolerate general anesthesia.
3. The perforating vessel is damaged -

Ages: 5 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: From April 2018 to August 2020, patients were hospitalized in the Department of Burns and Plastic Surgery of a regional hospital. All damages referred to the lower leg and soft tissue defects
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
flaps observation | 12-24months
  flaps color ,temperature ,with or without effusion

CONTACTS AND LOCATIONS:
Overall Officials: the affiliated hospital of xuzhou medical university, Study Chair — The Affiliated Hospital of Xuzhou Medical University
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choi JW, Nam SY, Choi SH, Roh JL, Kim SY, Hong JP. Applications of medial sural perforator free flap for head and neck reconstructions. J Reconstr Microsurg. 2013 Sep;29(7):437-42. doi: 10.1055/s-0033-1343959. Epub 2013 Apr 24. PMID 23616252
- [Background] Mendieta M, Cabrera R, Siu A, Altamirano R, Gutierrez S. Perforator Propeller Flaps for the Coverage of Middle and Distal Leg Soft-tissue Defects. Plast Reconstr Surg Glob Open. 2018 May 2;6(5):e1759. doi: 10.1097/GOX.0000000000001759. eCollection 2018 May. PMID 29922552